CLINICAL TRIAL: NCT03833830
Title: A Cross Sectional Study Assessing the Perifoveal and Peripapillar Vessel Density in nAMD After Longterm Anti-VEGF Treatment Compared to Recently Started Anti-VEGF Treatment - Pilotstudy
Brief Title: Vessel Density in nAMD After Longterm Anti-VEGF Treatment Compared to Recently Started Anti-VEGF Treatment
Status: Completed | Type: Observational
Sponsor: Dr. med. Katja Hatz (Other)
Collaborators: Cenaug Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Dr. med. Katja Hatz, Head of medical retina department, Vista Klinik
Organization: Vista Klinik (Other)
Other Study IDs: OCTA 2018-02043
Record Dates: First submitted 2018-12-27; First posted 2019-02-07 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- longterm treatment group: previous treatment (before Optical Coherence Tomography angiography (OCTA)) >20 injections
  Interventions: Diagnostic Test: Optical Coherence Tomography angiography (OCTA)
- shortterm treatment group: previous treatment (before Optical Coherence Tomography angiography (OCTA)) < 5 injections
  Interventions: Diagnostic Test: Optical Coherence Tomography angiography (OCTA)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography angiography (OCTA) — There will be an OCTA measurement (observational study) for both groups. Group allocation will be made due to previous anti-VEGF treatments (longterm treatment group >20 injections and shortterm treatment group < 5 injections).

SUMMARY:
Neovascular age-related macular degeneration (nAMD) is characterized by the abnormal growth of blood vessels from the choroid into the subretinal space which leads to sub- and intraretinal fluid accumulation, hemorrhages and subretinal fibrosis with progressive loss of central vision. Intravitreal anti-VEGF treatment is the standard of care. Intravitreal anti-VEGF application might temporarily increase intraocular pressure due to a volume effect. It remains unclear if repeated injections might have an impact on retinal capillary perfusion. Therefore this study aims to investigate the vascular microcirculation differences between patients who received longterm intravitreal Anti-VEGF treatment and patients who recently started Anti-VEGF treatment using Optical Coherence tomography Angiography (OCTA).

DETAILED DESCRIPTION:
Main outcome parameters are:

* Vessel Perfusion Area (%) of central ETDRS subfields and peripapillar region as evaluated by OCTA (single measurement)
* Blood flux index(*) of central ETDRS subfields and peripapillar region as evaluated by OCTA (single measurement).
* Peripapillary and perifoveal retinal nerve fiber layer (RNFL) thickness (µm) as evaluated by OCT (single measurement)
* Intraocular pressure (IOP) (mmHg) (single measurement at study visit) and mean intraocular pressure during anti-VEGF treatment period (evaluated as mean of all retrospectively available IOP measures from the beginning of treatment, mmHg)

(*)Blood flux index is automatically calculated by ARI Network as the mean flow intensity in the vessel area, where the blood flow signal was normalized to 0 to 1 by dividing by the full dynamic range of blood flow signal intensity.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation, patients will be required to

* have been treated for sub- or juxtafoveal CNV due to nAMD with anti-VEGF intravitreal injections either for at least 20 times (longterm treatment eyes) or <5 times (shortterm treatment eyes).
* give written consent to participation

Exclusion Criteria:

* diagnosis of glaucoma/ocular hypertension at baseline of anti-VEGF treatment

  * history of retinal vascular disorders like diabetic retinopathy, retinal vein/arterial occlusive disease, uveitis etc.
  * history of papillary disease which might interfere with interpretation of peripapillary OCT/OCTA evaluation such as severe tilted disc, parapapillar CNV, papillar drusen, optic nerve neuritis, papillar edema etc.
  * inability to perform OCTA examination of sufficient quality.
  * history of any side effects of Tropicamide eye drops

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive recruitment. All patients from Vista Klinik attending the retina outpatient clinic, who fulfil the in- and exclusion criteria, will be offered the participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Vessel Perfusion Area (%) and Flux index* of central ETDRS subfields and peripapillary region (single measurements at study visit), respectively, in both groups | baseline V0
  in both groups (longterm treatment group ( ≥20 intravitreal injections) and shortterm treatment group (<5 intravitreal injections).

SECONDARY OUTCOMES:
Peripapillary and perifoveal retinal nerve fiber layer (RNFL) thickness (µm) as evaluated by OCT (single measurement at study visit) | baseline V0
  in both groups (longterm treatment group ( ≥20 intravitreal injections) and shortterm treatment group (<5 intravitreal injections).
Intraocular pressure (IOP) (mmHg) (single measurement at study visit) and mean intraocular pressure during anti-VEGF treatment period (evaluated as mean of all retrospectively available IOP measures from the beginning of treatment, mmHg) | baseline V0
  in both groups (longterm treatment group ( ≥20 intravitreal injections) and shortterm treatment group (<5 intravitreal injections).
weight | baseline V0
  weight meassurements in kg
height | baseline V0
  height meassurements in cm

CONTACTS AND LOCATIONS:
Overall Officials: Katja Hatz, MD, Principal Investigator — Vista Klinik Binningen
Locations (1):
- Vista Klinik, Binningen, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
if necessary on request